CLINICAL TRIAL: NCT06894329
Title: Clinical Utility Study to Determine Impact of PanCystPro Assay on Physician Decision-making in the Management of Pancreatic Cystic Lesions
Brief Title: A Study for the PanCystPro Assay in the Management of Pancreatic Cystic Lesions
Acronym: PanAMP
Status: Not yet recruiting | Type: Observational
Sponsor: Amplified Sciences Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: PanAMP study
Record Dates: First submitted 2025-03-19; First posted 2025-03-25 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Pancreatic Cystic Lesions

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this research is to learn if the PanCystPro assay can help doctors in making decisions about treatment and monitoring of pancreatic cysts. The PanCystPro test measures glucose, carcinoembryonic antigen (CEA), and gastricsin biomarkers on fluid obtained from a pancreatic cyst. The test reports if the cyst fluid should be considered "Non-mucinous" or "Mucinous". Mucinous pancreatic cysts are more likely to progress to cancer while non-mucinous cysts seldom progress to cancer.

DETAILED DESCRIPTION:
A prospective observational study to assess the impact of PanCystPro in patients with radiographically confirmed pancreatic cysts planned for Endoscopic Ultra Sound (EUS) Fine Needle Aspirate (FNA). Eligible subjects will be enrolled after signing the ICF. One pancreatic cyst sample will be sent to the Amplified lab for PanCystPro testing.

The impact of PanCystPro on clinical management intention will be assessed after the PanCystPro result has been received by the physician. One year after enrollment the actual clinical management the patient received will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* Cross sectional imaging studies demonstrating a pancreatic cyst at least 12 mm in size where fluid sampling can aid in patient's management
* Written informed consent.
* The patient will be undergoing EUS with anticipated FNA extraction as part of standard patient care.

Exclusion Criteria:

* Patients diagnosed with pancreatic cancer.
* Pregnant or lactating females.
* Patients with contraindications to moderate or deep procedural sedation (necessary for the conduct of the endoscopic ultrasound) like major cardiorespiratory illness.
* Patients with contraindications to FNA of a pancreatic cyst like being on blood thinners.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with radiographically confirmed pancreatic cysts planned for EUS-FNA.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-06-15 (Estimated); Study Completion 2027-03-16 (Estimated)

PRIMARY OUTCOMES:
The percentage of subjects for which the providers indicated positive impact of the PanCystPro assay. | 1 month.
  The percentage of subjects for which the providers indicated positive impact on patient management decisions of the PanCystPro assay results in patients with radiographically confirmed pancreatic cysts.